CLINICAL TRIAL: NCT02706743
Title: Effect of Radioiodine Remnant Ablation on Quality of Life in Patients With Differentiated Thyroid Cancer:a Prospective Cohort Study
Brief Title: Assessment of Quality of Life After Adjunct Radioiodine Therapy in Patients With Differentiated Thyroid Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Sun Yungang, Principal Investigator, Southern Medical University, China
Other Study IDs: ZMing
Record Dates: First submitted 2015-05-29; First posted 2016-03-11 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Thyroid Neoplasms
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The aim of this study was to assess the impact of adjuvant radioactive iodine therapy on the quality of life(QOL) in differentiated thyroid cancer patients and to identify independent factors affecting changes in the QOL.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed new diagnosis of differentiated thyroid cancer, recently treated by total thyroidectomy
* Must sign a consent form before treatment
* One year or more of follow-up after radioiodine ablation

Exclusion Criteria:

* Patients with follicular, Hürthle cell, poorly differentiated, medullary, or anaplastic thyroid carcinoma
* Pregnant or lactating women
* Patients that received adjuvant radioiodine treatment in the past
* Patients with other cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with differentiated thyroid cancer initially referred to adjuvant radioiodine treatment in nuclear medicine department, Zhujiang Hospital, Southern Medical University.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in patients with differentiated thyroid cancer from baseline Medical Outcome Study Short-Form 36(MOS SF-36) questionnaire at 12 months | baseline and 12 months
  The Medical Outcome Study Short-Form 36(MOS SF-36) is a short questionnaire with 36 items which measure eight multi-item variables: physical functioning (10 items), social functioning (two items), role limitations due to physical problems(four items), role limitations due to emotional problems (three items), mental health (five items), energy and vitality (four items), pain (two items), and general perception of health (five items). For each variable item scores are coded, summed, and transformed on to a scale from 0 (worst possible health state measured by the questionnaire) to 100 (best possible health state).
Change in patients with differentiated thyroid cancer from baseline Hospital Anxiety and Depression Scale at 12 months | baseline and 12 months
  The Hospital Anxiety and Depression Scale HADS is a self-rated screening questionnaire detecting mild degrees of anxiety and depression. It consists of 14 questions, seven for anxiety and seven for depression. Scores range from non-cases (0-7 score), borderline cases(8-10 score), definite cases (11-21 score).
Change in patients with differentiated thyroid cancer from baseline Brief Fatigue Inventory at 12 months | baseline and 12 months
  The instrument is used to quickly assess the severity of fatigue experienced by cancer patients, as well as its impact on their ability to function over the previous 24 h.The BFI consists of 9 items on a single page. Fatigue and its interference are measured on numeric scales from 0-10. There are three items asking subjects to describe their fatigue now, at its usual level, and at its worst level during the previous 24 hours, using extreme points "no fatigue" and "fatigue as bad as you can imagine." The next six items describe how much fatigue has interfered with aspects of their life during the previous 24 hours. Specifically, these items are general activity, mood, walking ability, normal work (both work outside the home and daily chores), relations with other people, and enjoyment of life. These interference scales range from "0" ("does not interfere") to "10" ("completely in terferes"). The global score for the BFI is calculated as the mean value of these 9 items.

CONTACTS AND LOCATIONS:
Overall Officials: Sun Y Gang, Master, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital,Southern Medical University, Guangzhou, Guangdong, China